CLINICAL TRIAL: NCT03585673
Title: A Phase II Trial of Docetaxel-polymeric Micelles(PM) Plus Oxaliplatin as a First-line Chemotherapy in Patients With Esophageal Squamous Cell Carcinoma
Brief Title: Docetaxel-polymeric Micelles(PM) and Oxaliplatin for Esophageal Carcinoma
Acronym: DOSE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sung Yong Oh (Other)
Responsible Party: Sponsor-Investigator, Sung Yong Oh, Principal Investigator, Dong-A University Hospital
Organization: Dong-A University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAUHIRB-18-041
Record Dates: First submitted 2018-07-01; First posted 2018-07-13 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Esophagus Squamous Cell Carcinoma (SCC); Metastatic Cancer
Keywords: esophageal cancer; metastatic; inoperable; relapsed
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Neoplasm Metastasis; Esophageal Neoplasms; Recurrence | interventions — Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Docetaxel-PM + Oxaliplatin D1,8 every 3weeks until progression
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Docetaxel-PM+Oxaliplatin (Experimental): * Docetaxel-PM 35mg/m2 D1, 8 I.V.
  * Oxaliplatin 120mg/m2 D1 I.V. Every 3 weeks till progression
  Interventions: Drug: Docetaxel-PM; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Docetaxel-PM — Docetaxel-PM 35mg/m2 intravenous over 1hour day1 and 8 every 3 weeks till progression
  Other Names: NANOXEL-M
Drug: Oxaliplatin — Oxaliplatin 120mg/m2 intravenous over 2 hour day 1 every 3 weeks till progression
  Other Names: NEXATIN

SUMMARY:
Esophageal or esophageal-gastric junction squamous cell cancer has dismal prognosis. And still no promising chemotherapeutic drugs is existed. In this study, The investigators wanted to look at the effects and safety of first line docetaxel-PM and oxaliplatin weekly administration chemotherapy for the participants with inoperable or metastatic esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
Few results directly study the combination of docetaxel and oxaliplatin in the squamous cell cancer of the esophagus, but some studies have shown that it is safe to In the phase II study for the patients with gastroesophageal junction adenocarcinoma, a prior study reported the efficacy and safety of the combination therapy of docetaxel 80mg/m2 and oxaliplatin 100mg/m2 every 3 weeks schedule. Entire response rate was 34% and median survival duration was 11.6 months. Over grades 3 anemia and neutropenia were found in 17%, respectively, and non-hematological toxicities were mostly mild to moderate. In this study, a five-day preventive granulocyte colony-stimulating factor (G-CSF) was used to reduce hematology toxicity.

Meanwhile, there was the phase I/II studies of added capecitabine to docetaxel and oxaliplatin with divided schedule d1 and d8 every 3weeks for reducing toxicities. The subjects who participated in this study had at least one previous history of chemotherapy, but overall response rates were 43% and median values for the entire duration of survival were 9.8months. However, the side effects were significant, with 30 % of patients seeing diarrhea of Grade 3 or higher and 17 % seeing infection of Grade 3 or higher (SAE) reported at 37 %.

Looking at the reasons and background for this, the effects of docetaxel on esophageal squamous cell cancer patients are already known, and weekly divided administration has also demonstrated a reasonable level of effectiveness and safety. In studies conducted on gastric and esophageal adenocarcinoma, the combination of docetaxel and oxaliplatin also showed reasonable levels of effects and side effects.

In this study, The investigators wanted to look at the effects and safety of first line docetaxel-PM and oxaliplatin weekly administration chemotherapy for the participants with inoperable or metastatic esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. A patient whose squamous cell cancer of the esophagus or esophago-gastric junction has been confirmed by biopsy or cytology.
2. A patient who is not subject to local treatment such as surgical excision or concurrent definitive chemoradiotherapy.
3. Metastatic or relapsed esophageal cancer patients who planned first line palliative treatment.
4. Patients' age over 18
5. Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0-2
6. Patient has measurable lesions with RECIST v1.1
7. Patients with appropriate organ functions, such as the following, within seven days prior to the start of a clinical trial

   * Proper bone marrow function (ANC ≥ 1500/uL, Platelets ≥ 100,000/uL and Hb 8/microliter(uL))
   * Proper kidney function (serum creatinine ≤ 1.5 mg/L, 24-hour urine test or creatinine clearance ≥ 60 ml/min based on Cockcroft-Gault formula)
   * Appropriate liver function (bilirubin ≤ 1.5 mg/dL, transaminases aspartate transaminase (AST or SGOT) and alanine transaminase (AST or SGOT) ≤ 2.5 times normal upper limit)
8. Patients with at least three months of an expected life.
9. Signing written consent from patients or their legal guardians and understanding the right to withdraw consent at any time without disadvantage.

Exclusion Criteria:

1. In the case that the following treatment has been received in the past for the local stage treatment more than 6 months from the end of the treatment, enrolment is allowed.

   * Neoadjuvant chemotherapy
   * Concurrent or sequential chemoradiotherapy
   * Adjuvant chemotherapy
   * Adjuvant concurrent or sequential chemoradiotherapy
   * Definitive concurrent or sequential chemoradiotherapy
2. Patients with a history of administration of docetaxel, paclitaxel, or oxaliplatin at any time in the past.
3. Patients who have been treated for other active cancers other than esophageal cancer less than five years (but cured kin basal cell cancer or cured cervical carcinoma in situ are excluded).
4. The clinically confirmed esophagus obstruction, gastrointestinal bleeding, or perforation (except if the symptoms are sufficiently controlled through proper procedures such as stents).
5. Patients with significant, uncontrolled cardiovascular disease, infection, or infectious fever.
6. Patients with uncontrolled brain metastasis.
7. In the case of major surgery within the first two weeks of clinical trial treatment, the patient must recover sufficiently from the effects of this surgery.
8. Patients with pregnancy, breast feeding, or future plans.
9. Because of uncontrolled diabetes or diabetic neuropathy, patients who have any subjective symptoms regardless of their degree
10. Patients who have taken antihistamine or steroid within four weeks of clinical trial treatment
11. In combination with the state of Docetaxel-PM, patients who are not permitted to take combined medication (patients with severe renal dysfunction, para-platin, platinum compound, patients who have hypersensitivity to mannitol, etc.)
12. Patients with hypersensitivity history of Polysorbate 80
13. A patient who has hypersensitivity history to Docetaxel-PM or oxaliplatin or any drug containing platinum.
14. Patients with peripheral sensory neuropathy with functional impairment (may aggravate peripheral neuropathy) prior to clinical trial
15. Other cases

    * Have experienced an infection or other serious medical problems that could cause damage to a patient's functions, making it difficult for the patient to receive treatment in a research plan.
    * Mental, neurological, or dementia that can prevent a person from understanding and submitting a written statement and consent form
    * Patients who are certain to be out of the clinical trial or who cannot be monitored regularly for the following reasons: For example, psychological, social, family or geographical reasons, or conditions that make it difficult to observe or comply with appropriate clinical trial plans.
    * Uncontrolled hepatitis and chronic liver disease
    * Other patients who are judged unfit for clinical trials by their physicians and researchers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | up to 6 months
  complete response + partial response by RECIST

SECONDARY OUTCOMES:
Progression free survival | up to 12 months
  progression or death
Overall survival | up to 12 months
  death event
Adverse event | up tp 12 months
  Hypersensitivity or any side effects by NCI-Common Terminology Criteria for Adverse Events (CTCAE) v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Sung Yong Oh, MD, Principal Investigator — Dong-A University Hospital
Locations (1):
- Dong-A University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No